CLINICAL TRIAL: NCT05710757
Title: Investigating Proximal Muscle Strength Effects by Incorporating Proximal Muscle Lengthening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, LaToya Green, Associate Professor, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-08926-XP
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Proximal Muscle Strength; Proximal Muscle Lengthening
Keywords: blood flow restriction; myofascial release
MeSH Terms: interventions — Myofascial Release Therapy; Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: The control group will receive a sham myofascial release pectoralis minor release intervention. The experimental group will receive a myofascial release pectoralis minor release intervention. Both groups will receive blood flow restriction exercise to strength the scapula retractors.
Who Masked: Participant
Masking Description: The control group will receive a sham intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Myofascial Release (Experimental): The Experimental group will receive a myofascial release pectoralis minor release intervention.
  Interventions: Other: myofascial release; Device: blood flow restriction
- Sham Myofascial Release (Sham Comparator): The Control group will receive a sham myofascial release pectoralis minor release intervention.
  Interventions: Device: blood flow restriction; Other: myofascial release

INTERVENTIONS:
Other: myofascial release — Myofascial release (MFR) is a technique that involves applying gentle sustained pressure into the myofascial connective tissue restrictions to eliminate pain and restore motion.
  Arms: Myofascial Release
Device: blood flow restriction — Blood flow restricted (BFR) exercise is the brief and non-continuous blockage of venous blood flow using a device that restricts the flow of blood while exercising. This technique is used to produce hypertrophy (muscle growth) and strength responses while exercising at a lighter load than traditionally required to produce a similar response.
Other: myofascial release — Sham MFR.
  Arms: Sham Myofascial Release

SUMMARY:
The purpose of this study is to assess strength gains of proximal musculature in the nondominant upper extremity after implementing blood flow restriction (BFR) and myofascial release (MFR) with the supplementation of whey protein.

DETAILED DESCRIPTION:
The purpose of this study is to assess strength gains of proximal musculature in the nondominant upper extremity after implementing blood flow restriction (BFR) and myofascial release (MFR) with the supplementation of whey protein. Blood flow restricted (BFR) exercise is the brief and non-continuous blockage of venous blood flow using a device that restricts the flow of blood while exercising. This technique is used to produce hypertrophy (muscle growth) and strength responses while exercising at a lighter load than traditionally required to produce a similar response. Myofascial release (MFR) is a technique that involves applying gentle sustained pressure into the myofascial connective tissue restrictions to eliminate pain and restore motion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the age of 18 and 30

Exclusion Criteria:

* Individuals with uncontrolled high blood pressure
* Individuals with sickle cell anemia, current pregnancy
* Individuals with a history of deep vein thrombosis
* Individuals with diabetes
* Individuals with active infection
* Individuals with less than normal range of motion or muscle strength
* Individuals with moderate to severe upper extremity injury in the past 12 months
* Individuals with a current diagnosis of cancer.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Scapular retraction strength | 8 weeks
  Assess scapular retraction strength with a dynamometer

SECONDARY OUTCOMES:
One repetition maximum (1RM) | 8 weeks
  maximum amount of weight that can be lifted one time for scapular retractors on a row machine

OTHER OUTCOMES:
Length for the pectoralis minor | 8 weeks
  Assess length of the pectoralis minor with a tape measure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No